CLINICAL TRIAL: NCT04922775
Title: The Application of Traditional Chinese Medicine Functional Reduction in Muscle Fatigue
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: China Medical University, Taiwan (Other)
Responsible Party: Principal Investigator, Han-Kuei Wu, Assistant Professor, China Medical University, Taiwan
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: TCM-Taping
Record Dates: First submitted 2021-06-01; First posted 2021-06-11 (Actual); Last update posted 2021-06-11 (Actual); Status verified 2021-06

CONDITIONS: Muscle Fatigue
Keywords: taping; Chinese medicine reduction; muscle fatigue

STUDY DESIGN:
Intervention Model Description: Participants will be categorized into two (A&B) groups randomly for cross-over study. A group will accept conventional taping before muscle fatigue exercise for the first course then accept Chinese medicine technique taping before muscle fatigue exercise for the second course. B group will accept Chinese medicine technique taping before muscle fatigue exercise for the first course then accept conventional technique taping before muscle fatigue exercise for the second course.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- conventional taping-Chinese medicine technique taping (Other): Participants will accept conventional taping before muscle fatigue exercise for the first course then accept Chinese medicine technique taping before muscle fatigue exercise for the second course.
  Interventions: Procedure: conventional taping; Procedure: Chinese medicine technique taping
- Chinese medicine technique taping-conventional taping (Other): Participants will accept Chinese medicine technique taping before muscle fatigue exercise for the first course then accept conventional technique taping before muscle fatigue exercise for the second course.
  Interventions: Procedure: conventional taping; Procedure: Chinese medicine technique taping

INTERVENTIONS:
Procedure: conventional taping — Participants will accept conventional taping before muscle fatigue exercise.
Procedure: Chinese medicine technique taping — Participants will accept Chinese medicine technique taping before muscle fatigue exercise.

SUMMARY:
In this study, 45 healthy participants between 20 and 40 of age will be included. After obtaining the consent, the participants will be categorized into two(A&B) groups randomly for cross-over study. Each of group will accept either conventional taping or Chinese medicine technique taping before muscle fatigue exercise. To compare the preventive effect, Myoton PRO, pulse analysis equipment, etc will be applied for evaluation. The application of Chinese medicine technique (ie. Chinese medicine functional reduction) taking the kinetic chain into consideration may improve body's functional movement.

DETAILED DESCRIPTION:
Nowadays, the importance of exercise is highly valued. The prevalence of sports injury is also increasing and may be associated with muscle fatigue. Therefore, the study focused on the prevention of common muscle fatigue in legs during exercise. With the modern sport medicine knowledge and kinesio taping, the investigators tried to figure out whether muscle fatigue can be diminished through the concept of Chinese medicine channel sinews techniques in advance. In this study, 45 healthy participants between 20 and 40 of age will be included. The exclusion criteria are as follows: i.pregnancy ii.current health problem iii.injuries of legs within a month. After obtaining the consent, the participants will be categorized into two(A&B) groups randomly for cross-over study. Each of group will accept either conventional taping or Chinese medicine technique taping before muscle fatigue exercise. To compare the preventive effect, Myoton PRO, pulse analysis equipment, etc will be applied for evaluation. The application of Chinese medicine technique (ie. Chinese medicine functional reduction) taking the kinetic chain into consideration may improve body's functional movement. Our goal is to enhance the coordination of the entire body structure, not merely the partial body structure improvement. In this way, it will benefit the prevention of exercise injuries and therapeutic effect.

ELIGIBILITY:
Inclusion Criteria:

* participants between 20 and 40 of age

Exclusion Criteria:

* i.pregnancy ii.current health problem iii.injuries of legs within a month

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2020-08-18 (Actual); Primary Completion 2020-12-26 (Actual); Study Completion 2020-12-26 (Actual)

PRIMARY OUTCOMES:
Muscle tone | one week
  The soft tissue will be evaluated by Myoton PRO. The muscle tone is measured by the "oscillation frequency (HZ)" characterizing the tone of a muscle in its passive or resting state without any voluntary contraction. Abnormally high muscle tine would slow the muscle recovery.
Muscle stiffness | one week
  The soft tissue will be evaluated by Myoton PRO. The muscle stiffness is evaluated by the "dynamic stiffness (N/m)" characterizing the resistance to a contraction or to an external force that deforms its initial shape. Abnormally high stiffness may lead to an inefficient economy of movement.
Muscle elasticity | one week
  The muscle elasticity is evaluated by the "logarithmic decrement" of a tissue's natural oscillation characterizing the ability to recover its initial shape after a contraction of removal an external force of deformation. If the decrement of a muscle decreases, the muscle elasticity increases.
Muscle relaxation | one week
  The muscle relaxation is evaluated by the "mechanical stress relaxation time (ms)" characterizing the time for a muscle to recover its shape from deformation after a voluntary contraction or a removal of an external force.
Muscle creep | one week
  The creep is evaluated by the "ratio of deformation and relaxation time" characterizing the gradual elongation of tissue over time when placed under a constant tensile stress.

SECONDARY OUTCOMES:
Pain scale | one week
  Pain assessment by the Wong-Baker Faces Pain Rating Scale. The scale shows a series of faces ranging from a happy face at 0, or "no hurt", to a crying face at 10, which represents "hurts like the worst pain imaginable".
Pulse wave | one week
  Radial pulse wave analysis

CONTACTS AND LOCATIONS:
Overall Officials: Chia-Hung Tien, Bachelor, Study Director — China Medical University, Taiwan
Locations (1):
- China Medical University, Taichung, Taiwan